CLINICAL TRIAL: NCT01563120
Title: A Comparison Between Two Oral Hypoglycemics - Metformin and Glybenclamide for the Treatment of Gestational Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0002-11-EMC
Record Dates: First submitted 2011-12-28; First posted 2012-03-26 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Glyburide

ARMS (2):
- metformin (Active Comparator): metformin up to 2550mg per day
  Interventions: Drug: metformin
- glybenclamide (Active Comparator): glybenclamide up to 20mg per day.
  Interventions: Drug: glybenclamide

INTERVENTIONS:
Drug: metformin — metformin up to 2550mg per day.
  Arms: metformin
Drug: glybenclamide — glybenclamide up to 20mg per day.
  Arms: glybenclamide

SUMMARY:
Rationale Gestational diabetes mellitus (GDM) complicates 5-7% of pregnancies. Major hazards include macrosomia, polyhydramnios, labor trauma and neonatal hypoglycemia. The ADA and ACOG recommend glucose control in order to reduce the incidence of hyperglycemia induced complications. Glucose control can be achieved using diet and life style changes. Insulin is initiated in women who fail to obtain glucose control with diet alone. During the past 11 years oral hypoglycemic drugs have been tested and proven to be efficacious and safe.

Objectives

1. To compare the efficacy and safety of glybenclamide vs. metformin in the treatment of women diagnosed with GDM
2. To evaluate the improvement in glycemic control after the addition of a second oral hypoglycemic drug after failure of the first

Hypothesis GDM is one of the major conditions contributing to obstetrical complications and prenatal morbidity. Improving glycemic control, by means of improving compliance and patient satisfaction, will decrease obstetrical complications, maternal and neonatal morbidity and have positive long term health implications.

Study design Prospective, randomized, open label

Study population Women between the ages 18-45, diagnosed with GDM will be recruited. GDM will be defined by a pathological OGTT (according to Carpenter and Coustan criteria) performed at or after 13 weeks of gestation.

Study period From recruitment until discharge of the newborn baby after delivery

Study protocol Women will be randomized at recruitment. Demographic and obstetrical data will be collected. Average glucose levels during the previous two weeks, estimated fetal weight and amniotic fluid index, and lab exams reflecting glycemic control will be noted. Women will provide daily glucose levels via fax or mail once a week. Glycemic control will be evaluated by a daily chart, including 7 measurements: 3 preprandial, 3 postprandial and a 7th measurement at 10 pm. Women will be invited to a monthly follow-up, which will include a sonographic evaluation of fetal weight and amniotic fluid, and lab exams. Follow-up protocol after 38 w of gestation will be according to our ward's protocol. The study was approved by the local Helsinki committee.

Time table Duration: two years

ELIGIBILITY:
Inclusion Criteria:

1. Patients with GDM with a gestational age between 14-33 weeks
2. Fasting glucose over 95 mg% or over 130 mg% an hour and a half postprandial (PPD) or a daily average over 100 mg%
3. At least a week of dietary treatment
4. Sonographic dating of the pregnancy earlier than 24 weeks
5. Signing a consent form

Exclusion Criteria:

1. Suspected IUGR earlier than 24 week of gestation
2. Major fetal malformation
3. Pre-gestational diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
glycemic control | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. OB/GYN, Emek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Nachum Z, Zafran N, Salim R, Hissin N, Hasanein J, Gam Ze Letova Y, Suleiman A, Yefet E. Glyburide Versus Metformin and Their Combination for the Treatment of Gestational Diabetes Mellitus: A Randomized Controlled Study. Diabetes Care. 2017 Mar;40(3):332-337. doi: 10.2337/dc16-2307. Epub 2017 Jan 11. PMID 28077460